CLINICAL TRIAL: NCT03483922
Title: Clinical Trials on Detection of Hepatocellular Carcinoma With Non-invasive Method Based on DNA Methylation of Circulated Tumor DNA, PBMC and T Cells
Brief Title: HCC Screening Using DNA Methylation Changes in ctDNA
Status: Completed | Type: Observational
Sponsor: HKGepitherapeutics (Industry)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Other Study IDs: HKG-Bng-HCC-100
Record Dates: First submitted 2018-03-20; First posted 2018-03-30 (Actual); Results first posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood monocyte (PBMC) DNA and plasma free circulating DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- chronic hepatitis B: This group will include 50 with hepatitis B subjects and the diagnoses will be based on AASLD practice guideline.
  Interventions: Diagnostic Test: ctDNA methylation in and it's Correlation wth Development and prediction of HCC
- HCC Cases: This group will include 350 in stage 0, stage A, stage B, Stage C+D of hepatocellular carcinoma.
  HCC staging will be diagnosed according to EASL-EORTC Clinical Practice Guidelines: Management of hepatocellular carcinoma
  Interventions: Diagnostic Test: ctDNA methylation in and it's Correlation wth Development and prediction of HCC
- Healthy: This group will include 50 healthy sex and age matched controls.
  Interventions: Diagnostic Test: ctDNA methylation in and it's Correlation wth Development and prediction of HCC

INTERVENTIONS:
Diagnostic Test: ctDNA methylation in and it's Correlation wth Development and prediction of HCC — Blood sample from patients with HCC, healthy individuals and individuals with hepatitis B will be collected, and DNA will extracted from PBMC and circulated tumor DNA will be subjected to bisulfite conversion. DNA from PBMC DNA will be analyzed with primers developed for the AHNAK-STAP1 genes. Plasma samples will be subjected to EZ direct DNA extraction and bisulfite conversion kit and will be amplified with primers developed to amplify the target regions. DNA will be used for the subsequent PCR amplification with specific primer to generate PCR amplicon for sequencing using a double PCR procedure. The product of PCR reaction will be subjected to indexed MiSeq Next-Generation sequencing that will allow us quantify DNA methylation level.

SUMMARY:
Hepatocellular Carcinoma (HCC) is the fifth most common cancer world-wide. It is particularly prevalent in Asia, and its occurrence is highest in areas where hepatitis B is prevalent, indicating a possible causal relationship. Follow up of high-risk populations such as chronic hepatitis patients and early diagnosis of transitions from chronic hepatitis to HCC would improve cure rates. In most cases HCC is detected late resulting in increased mortality and morbidity.

The purpose of this study is to develop and test non-invasive biomarkers based on methylation changes in PBMC and circulated tumor DNA in hepatocellular carcinomas patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC by EASL-EORTC guidelines
* Confirmed hepatitis B diagnosis for HepB patients using AASLD practice guidelines.

Exclusion Criteria for HCC:

* Cirrhosis, any other known inflammatory disease (bacterial or viral infection with the exception of hepatitis B or C, diabetes, asthma, autoimmune disease, active thyroid disease) which could alter T cells and monocytes characteristics
* Other cancers.

Exclusion Criteria for HepB:

* Diagnosis of HCC or any other cancer.

Exclusion Criteria for Healthy Controls:

* Any known inflammatory or infectious disease including HepB and HepC
* Chronic diseases,
* Cancer
* Medications or drug use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC staging will be diagnosed according to EASL-EORTC Clinical Practice Guidelines: Management of hepatocellular carcinoma. The patients will be divided into four groups, including Stage 0 (1) (n=100), stage A (2) (n=100), stage B (3) (n=100) and stage C+D (4) (n=100). As controls we will recruit chronic hepatitis B (n=100), which diagnose will be confirmed using AASLD practice guideline for chronic Hepatitis B, and healthy sex and age matched controls (n=100).
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Ali Khan, PhD, Principal Investigator — nternational Centre for Diarrhoeal Disease Research
Locations (1):
- Infectious Diseases Division, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy: This group included 49 healthy sex and age matched controls.
- Chronic Hepatitis B: This group included 51 Chronic hepatitis B patients
- HCC Stage 0: This group included two patients with stage 0 (very early stage)
- HCC Stage A: This group included 32 patients with stage A (early stage)
- HCC Stage B: This group included 86 patients with stage B (intermediate stage) of HCC
- HCC Stage C: This group included 106 patients with stage C (advanced stage) of HCC
- HCC Stage D: This group included 76 patients with stage D (end stage) of HCC
Period: Overall Study
Arm/Group | Healthy | Chronic Hepatitis B | HCC Stage 0 | HCC Stage A | HCC Stage B | HCC Stage C | HCC Stage D
Started | 49 | 51 | 2 | 32 | 86 | 106 | 76
Completed | 49 | 51 | 2 | 32 | 86 | 106 | 76
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 402 participants were recruited from the Dhaka area to the study included 49 healthy controls, 51 Chronic hepatitis B patients and 302 HCC patients from stages 0 to D (HCC O n=2, HCCA n=32, HCC B n=86, HCC C n=106, HCC D n=76)
Groups:
- Healthy: Healthy controls
- Chronic Hepatitis B: Chronic hepatitis B patients
- HCC Stage 0: HCC patients with Stage 0
- HCC Stage A: HCC patients with Stage A
- HCC Stage B: HCC patients with Stage B
- HCC Stage C: HCC patients with Stage C
- HCC Stage D: HCC patients with Stage D
- Total: Total of all reporting groups
Arm/Group | Healthy | Chronic Hepatitis B | HCC Stage 0 | HCC Stage A | HCC Stage B | HCC Stage C | HCC Stage D | Total
Number analyzed (Participants) | 49 | 51 | 2 | 32 | 86 | 106 | 76 | 402
Age, Continuous [Mean (Full Range); unit: years] | 26.14 [18 to 47] | 28.71 [18 to 46] | 62 [57 to 67] | 49.15 [19 to 67] | 49.12 [18 to 70] | 49.34 [18 to 70] | 52.45 [25 to 70] | 44 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 0 | 5 | 14 | 21 | 12 | 68
  Male | 42 | 42 | 2 | 27 | 72 | 85 | 64 | 334
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 49 | 51 | 2 | 32 | 86 | 106 | 76 | 402
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Bangladesh | 49 | 51 | 2 | 32 | 86 | 106 | 76 | 402

OUTCOME MEASURES:

1. Primary Outcome: Calculation of M Scores and HCC Probability Scores
Description: We normalized median methylation values (range 0-100) for 'HCC-detect' (Hepatocellular Carcinoma Detection) and 'HCC-spec' (Hepatocellular Carcinoma Specificity). 'HCC-detect' is derived from CHFR, VASH2, CCNJ, and GRID2IP regions, aiming to broadly identify HCC. Theoretical range is -6.6438 to 8.6438, with observed -3.541 to 7.65; higher scores indicate increased HCC likelihood. 'HCC-spec', focusing on the F12 region, differentiates HCC from 31 other cancers and normal cells, with theoretical range -3.3219 to 6.64385 (observed -3.3219 to 6.6297). Higher scores signify greater HCC specificity. Both scores, modeled via logistic regression in Prism, predict HCC probability, linking higher scores with higher HCC likelihood or specificity
Time Frame: 6 months to 1 year
Population: Out of the 402 participants, five did not meet the sequencing depth threshold (i.e., less than 100 reads per gene) for at least one gene, and they were excluded from subsequent analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Chronic Hepatitis B: Patients with chronic hepatitis B
- HCC Stage 0: Patients with stage 0 HCC
- HCC Stage A: Patients with stage A HCC
- HCC Stage B: Patients with stage B HCC
- HCC Stage C: Patients with stage C HCC
- HCC Stage D: Patients with stage D HCC
Arm/Group | Healthy | Chronic Hepatitis B | HCC Stage 0 | HCC Stage A | HCC Stage B | HCC Stage C | HCC Stage D
Number analyzed (Participants) | 46 | 49 | 2 | 32 | 86 | 106 | 76
units on a scale | 1.113 (0.3267) | 1.159 (0.3508) | 1.797 (0.2483) | 1.707 (0.3615) | 1.839 (0.2268) | 1.818 (0.2525) | 1.891 (0.215)

ADVERSE EVENTS:
Time Frame: Our observational study, focused on identifying biomarkers for HCC detection, did not involve the collection or monitoring of adverse event data. The duration for participant involvement spanned from the study start date of August 20, 2018, to the primary completion date of June 1, 2020. During this period, spanning approximately 1 year and 9 months, there were 0 participants at risk for adverse events due to the non-interventional nature of the study.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored or assessed because the study was non-interventional and focused solely on testing liquid biopsy methylation markers. Therefore, no participants were at risk for adverse events.
Groups:
- Healthy: 49 healthy controls
- Chronic Hepatitis B: 51 Chronic hepatitis B patients
- HCC Stage 0: 2 patients with stage 0 of HCC
- HCC Stage A: 32 patients with stage A of HCC
- HCC Stage B: 86 patients with stage B of HCC
- HCC Stage C: 106 patients with stage C of HCC
- HCC Stage D: 76 patients with stage D of HCC
Arm/Group | Healthy | Chronic Hepatitis B | HCC Stage 0 | HCC Stage A | HCC Stage B | HCC Stage C | HCC Stage D
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Inherent challenges of our study included a regional focus and a reliance on observational data, which may limit broader applicability and prevent establishing causal relationships. Technical aspects, like the exclusion of participants due to insufficient sequencing depth (less than 100 reads per gene for five out of 402 participants), reflect constraints in data robustness. These elements represent areas for potential enhancement in future research

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03483922/Prot_SAP_000.pdf